CLINICAL TRIAL: NCT01835405
Title: A Prospective, Single-centre Study to Compare the Use of LiquiBand® Flex, Dermabond Advanced™ or Conventional Sutures for the Topical Closure of Surgical Wounds
Brief Title: LiquiBand Versus Dermabond Versus Sutures for Closure of Surgical Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-LBF001-05-1
Record Dates: First submitted 2013-04-12; First posted 2013-04-19 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Surgical Incisions
MeSH Terms: conditions — Surgical Wound | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- LiquiBand Flex (Active Comparator): LiquiBand® Flex skin adhesive is indicated for topical application only, to hold closed easily approximated skin edges from surgical incisions, including punctures from minimally invasive surgery, and simple, thoroughly cleansed trauma-induced lacerations. It may be used in conjunction with, but not in place of deep dermal sutures.
  Interventions: Device: LiquiBand Flex
- Dermabond Advanced (Active Comparator): Dermabond Advanced™ adhesive is intended for topical application only, to hold closed easily approximated skin edges of wounds from surgical incisions, including incisions from minimally invasive surgery, and simple, thoroughly cleansed, trauma-induced lacerations. Dermabond Advanced ™ adhesive may be used in conjunction with, but not in place of, deep dermal stitches.
  Interventions: Device: Dermabond Advanced
- Sutures (Prolene) (Active Comparator): Prolene™ Suture is indicated for use in general soft tissue approximation and/or ligation, including use in cardiovascular, ophthalmic and neurological procedures.
  Interventions: Device: Sutures (Prolene)

INTERVENTIONS:
Device: LiquiBand Flex
  Arms: LiquiBand Flex
Device: Dermabond Advanced
  Arms: Dermabond Advanced
Device: Sutures (Prolene)
  Arms: Sutures (Prolene)

SUMMARY:
To evaluate the cosmetic outcome, effectiveness, user and subject satisfaction, and safety of LiquiBand® Flex in relation to DermaBond Advanced™ and conventional sutures for the topical closure of surgical wounds.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 or older on day of enrollment
* Scheduled for surgical procedure by a delegated study surgeon
* Fresh surgical wound with evenly distributed tension over length of incision
* Willing and able to sign informed consent
* Agree to return for 2 week (+/- 7 days) and 3 month (90 days +/- 7 days) post-procedure follow-up visit

Exclusion Criteria:

* Known sensitivity to cyanoacrylates, formaldehyde or acetone products
* Wounds in which incision edges are under high tension or not easily apposed (after deep layer suture), or over joints (unless immobilized)
* Wounds less than 15mm in length
* Wounds in which haemostasis is not able to be achieved, eg, drain is placed or Warfarin level >2.5 prior to surgery
* Wounds in which deep closure could not be achieved
* Surgical procedures involving mucus membranes or eyes
* Mental incapacity, dementia, or inability to give informed consent
* Pregnant or nursing
* Disease related or pharmacologically immuno-compromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2014-02-14 (Actual); Study Completion 2014-02-14 (Actual)

PRIMARY OUTCOMES:
To compare cosmetic outcomes at follow up | 3 months post treatment
  Cosmesis to be evaluated by a panel of masked evaluators using a modified Hollander Wound Evaluation Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Care Center, Beverly Hospital, Beverly, Massachusetts, United States